CLINICAL TRIAL: NCT05779202
Title: Observational Study on Cardiac Biomarkers Testing in Patients with Muscular Dystrophy Cardiomyopathy and Assessing the Feasibility of Serial Cardiac Troponin Testing At 0 Hour and 1 Hour, As Well As the Mid-term Biovariability of Cardiac Troponin
Brief Title: Observational Study on Cardiac Biomarkers Testing in Patients with Muscular Dystrophy Cardiomyopathy
Acronym: KYMA
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mustafa Yildirim, Principal Investigator, University Hospital Heidelberg
Other Study IDs: KYMA
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathies; Skeletal Muscle Disorder
MeSH Terms: conditions — Cardiomyopathies; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Routine blood samples at presentation, a second blood sample for study purposes will be collected after 1 hour of the first index visit. On the routine follow-up visit, we will collect 20 ml for storage in addition to the routine blood test. Blood samples will be obtained by standard venous blood sampling. Assessment of parameters include laboratory values with special focus on findings related to myocardial injury as indicated by high sensitivity cardiac troponin T (hs-cTnT) and hs-cTnI. Moreover, the laboratory panel comprises other cardiac biomarkers, electrolytes, renal (creatine, glomerular filtration rate) and liver function (GOT, GPT, LDH), C-reactive protein, D-dimer etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention is planned. — No intervention is planned.

SUMMARY:
The objective of this study is to evaluate acute changes of cardiac troponin (and other cardiac biomarkers) and mid-term biovariability in patients with cardiomyopathy associated with chronic skeletal muscle disease. The specific aims of the study are:

Firstly, to evaluate the feasibility of the ESC 0/1 hour protocol for rule-in and rule-out of a non-ST-segment elevation acute coronary syndrome (NSTE-ACS).

Secondly, a) to determine reference change values (RCV) to characterize physiological biovariability, b) to differentiate acute from chronic high-sensitivity cardiac troponin T (hs-cTnT) elevations.

DETAILED DESCRIPTION:
In patients with skeletal muscle dystrophy, cardiac involvement is one of the limiting factors regarding mortality. Early detection of a dystrophy-associated cardiomyopathy is important, as heart failure therapy can slow adverse cardiac remodeling and alleviate heart failure symptoms. Cardiac biomarkers, especially high-sensitivity cardiac Troponin T (hs-cTnT) and to a lesser extent, high-sensitivity cardiac Troponin I (hs-cTnI), are chronically elevated in diseases with underlying structural heart disease. However, there is no reliable data on whether changes in the concentration of cardiac Troponin T or I are suitable for monitoring the cardiac disease progression. This can lead to delayed diagnosis and treatment of a relevant deterioration of the disease or even acute heart muscle damage in the context of acute myocardial infarction, pulmonary embolism, and myocarditis. Due to insufficient clinical data, the feasibility and safety of the ESC 0/1-hour protocol according to the ESC guidelines for the diagnosis of acute myocardial infarction in this patient population are uncertain. Furthermore, it is necessary to determine the normal biovariability of high-sensitivity cardiac Troponin T (hs-cTnT) and high-sensitivity cardiac Troponin I (hs-cTnI) to differentiate physiological concentration fluctuations of these cardiac biomarkers in this patient population from changes that represent an improvement or deterioration of heart function. Routine blood samples that will be collected at presentation, a second blood sample for study purposes will be collected after 1 hour for the first index visit. On the routine follow-up visit, 20 ml of blood will be collected for storage in addition to the routine blood test. Blood samples will be obtained by standard venous blood sampling. If venipuncture is unsuccessful or considered harmful by the patient and a suitable peripheral venous catheter is available, the venous catheter may be used for blood sampling to minimize damage. Assessment of parameters includes demographics and clinical characteristics (symptoms, history, medication, vital signs, risk scores etc.) and laboratory values with special focus on findings related to myocardial injury as indicated by high sensitivity cardiac troponin T (hs-cTnT) and hs-cTnI. Moreover, the laboratory panel comprises other cardiac biomarkers, electrolytes, renal (creatine, glomerular filtration rate) and liver function (GOT, GPT, LDH), C-reactive protein, D-dimer etc.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosed muscular dystrophy
* Patients >18 years of age

Exclusion Criteria:

* Patients with poor venous status
* Hemodialysis
* Lack of capacity to provide informed consent or refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with cardiomyopathy associated with chronic skeletal muscle disease presenting at Heidelberg University Hospital in the cardiomyopathy outpatients' clinic during a time period of 12 months are eligible for study inclusion.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of stable troponin kinetics in patients | 1 hour
  The first main objective is to determine the prevalence of stable troponin kinetics defined as high-sensitivity Troponin T (hour 0) : high-sensitivity Troponin T (hour 1) < 5 ng/l at baseline presentation.
Reference Change Values calculation for cardiac biomarkers | 6 months
  The second main objective is to calculate the Reference Change Values (RCV) of high-sensitivity Troponin T within the 6-month follow-up period.

SECONDARY OUTCOMES:
Longitudinal follow-up of novel laboratory biomarkers for prognostic significance. | unlimited
  Thirdly, longitudinal follow-up of the patients will be conducted once a year to clarify the prognostic significance of novel laboratory biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No